CLINICAL TRIAL: NCT03770052
Title: A Double Blind, Randomized, Investigator Initiated Study on Glucose-Lowering Effects and Safety of Adding 0.25 or 0.5 mg Duvie (Lobeglitazone) in Patients With Type 2 Diabetes With Inadequate Control on Metformin and DPP-4 Inhibitor Therapy
Brief Title: Glucose-Lowering Effects and Safety of Adding 0.25 or 0.5 mg Duvie
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Principal Investigator, In Ju Kim, Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Duvie2.5
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes Mellitus; Inadequate Glucose Control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.25mg robeglitazone add-on group (Experimental): 0.25mg robeglitazone once daily in patients with type 2 diabetes with inadequate control on metformin and DPP-4 inhibitor therapy
  Interventions: Drug: duvie
- 0.5mg robeglitazone add-on group (Active Comparator): 0.5mg robeglitazone once daily in patients with type 2 diabetes with inadequate control on metformin and DPP-4 inhibitor therapy
  Interventions: Drug: duvie

INTERVENTIONS:
Drug: duvie — take the intervention drug once daily according to the randomized groups

SUMMARY:
Glucose-Lowering Effects and Safety of Adding 0.25 or 0.5 mg Duvie

DETAILED DESCRIPTION:
This study is a double blind, randomized, investigator initiated study on glucose-lowering effects and Safety of Adding 0.25 or 0.5 mg Duvie (Lobeglitazone) in Patients With Type 2 Diabetes With Inadequate Control on Metformin and DPP-4 Inhibitor Therapy. The primary aim of the study is to compared changes of HbA1c between 0.25mg robeblitazone add-on group and 0.5mg robeglitazone add-on group.

ELIGIBILITY:
Inclusion Criteria:

1. Type Ⅱ diabetes mellitus
2. Between 19 years and 80 years old
3. BMI between 20kg/㎡ to 45kg/㎡
4. Among those using Metformin and DPP-4 inhibitor merging therapy for more than 3 months, A person who has not changed the dosage of Metformin 500 mg and DPP-4 inhibitor for more than 8 weeks at the time of screening
5. HbA1c 7.0 to 9.0
6. Agreement with written informed consent

Exclusion Criteria:

1. Historical history of severe heart failure or heart failure (NYHA Class III&IV)
2. Rapid coronary syndrome, cardiovascular interventions within 6 months
3. History of cerebral vascular diseases within six months
4. High blood pressure uncontrolled (>160/100 mmHg)
5. In case weight loss drug is used within 3 months
6. In case of systemic corticosteroids treatment within 3 months
7. If there is an allergy or overreaction to the study drug or its components
8. In case of acute metabolic complications (ketonicemia or high osmotic pressure) within 6 months
9. Anemia Hb < 12g/dL(male), 10g/dL(female)
10. Kidney function GFR < 45mL/min/1.73m2 (GFR test results are calculated by the Cockcroft-Gault Calculator).
11. impaired hepatic function (AST/ALT 2.5-fold the upper limit of the normal range [ULN])
12. TG>500 mg/dL
13. LDL cholesterol >160 mg/dL

    - If a lipid-lowering agent is being taken, the existing dose should be taken during the study period.
14. The thyroid hormone is within its normal range

    - however, thyroid hormone may be registered at the discretion of the investigator even if it is outside the normal range.
15. Laser treatment for proliferative retinopathy within 6 months
16. history of alcohol or drug abuse in the previous 3 months
17. history of most cancers not in remission for 5 years
18. Past history of bladder cancer
19. Women nursing or pregnant Persons who are not using effective contraceptive methods, or who refuse to use contraceptives as specified below (permitted contraceptives: condoms, castings, or implantation contraceptives, etc.) are installed with contraceptives in the uterus
20. external injury, acute infections, a history/presence of any other severe disease, or severe trauma
21. Patients who use basins - however, they can be registered by stopping 8 weeks before the start of administration of medicines for clinical trials
22. A person who has used endemic insulin for more than 7 days in the last 8 weeks
23. A person with the drug usage in the TZD series over the last eight weeks.
24. When experiencing allergies, hypersensitivity, or side effects associated with drug use in the TZD series;
25. The researcher determines that other participants may experience difficulties in participating in the test through to the end, or that participation in the test may result in additional risks or confusion in the test results.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
HbA1c at 24 week | 24 week
  changes of HbA1c between baseline and 24 week

SECONDARY OUTCOMES:
HOMA-IR | 24 week
  changes of HOMA-IR between baseline and 24 week
lipid levels | 24 week
  changes of lipid levels between baseline and 24 week
hs-CRP | 24 week
  changes of hs-CRP between baseline and 24 week
AST | 24 week
  changes of AST between baseline and 24 week
adiponectin | 24 week
  changes of adiponectin between baseline and 24 week
adverse event (weight gain,edema) | 24 week
  changes of adverse event (weight gain,edema) between baseline and 24 week
ALT | 24 week
  changes of ALT between baseline and 24 week
ALP | 24 week
  changes of ALP between baseline and 24 week
total bilirubin | 24 week
  changes of total bilirubin between baseline and 24 week

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No